CLINICAL TRIAL: NCT02422433
Title: Surveillance and Image-Guided Biopsy of the Esophagus Using an OFDI Capsule
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-P001254; 5R01CA103769-08 (NIH)
Record Dates: First submitted 2014-07-25; First posted 2015-04-21 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Barrett's Esophagus
Keywords: EGD; OFDI; Barrett's Esophagus; Imaging; Biopsy; OCT
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OFDI Capsule Marking and Imaging (Experimental): Participant will swallow the OFDI capsule, marking will be performed by making superficial cautery marks on the tissue. This will be followed by imaging using the OFDI Imaging system.
  Interventions: Device: OFDI Capsule Marking

INTERVENTIONS:
Device: OFDI Capsule Marking — Marking and imaging of the esophagus using the OFDI Capsule and system.

SUMMARY:
The purpose of this research is to test the feasibility, sensitivity, and specificity of the marking Optical Frequency Domain Imaging (OFDI) capsule for diagnosing Barrett's Esophagus (BE).

DETAILED DESCRIPTION:
A total of 130 participants scheduled to undergo esophagogastroduodenoscopy (EGD) will be asked to swallow the OFDI capsule while being unsedated. The capsule is attached to a tether that allows the capsule operator to navigate the capsule as it progresses down the esophagus using natural propulsion called peristalsis as well as to bring it back up to pulled out of the mouth when the procedure is done.

OFDI real-time images will be used for targeting of the region to be marked. Once in position, two cautery marks will be made to only the superficial layers of the esophageal mucosa. Following cautery marking, the capsule will be lowered in the esophagus and marked regions of interest will be reimaged for confirmation of the placement of potential cautery marks.

Immediately following the completion of the experimental procedure, the standard of care with the performance of the surveillance endoscopy will be performed. Images obtained by the OFDI capsule will be compared to the images obtained by the clinical endoscopy and histology.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be undergoing an EGD.
* Patients must be over the age of 18.
* Patients must be able to give informed consent.

Exclusion Criteria:

* Patients who are on anti-platelet medications or anti-coagulation medications, and NSAIDS at the time of procedure.
* OR patients with a history of hemostasis disorders.
* OR patients with esophageal strictures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the marking OFDI capsule for diagnosing BE by comparing OFDI images and biopsy diagnosis | It is expected that the total experimental time including swallowing the OFDI capsule OFDI, OFDI imaging, and removal of the OFDI capsule will take approximately 20 minutes
  The images obtained by the OFDI capsule will be compared to the images obtained by the clinical endoscopy and histology.

SECONDARY OUTCOMES:
Sensitivity of the marking OFDI Capsule to correctly detect and mark the region of interest in BE | It is expected that the total experimental time including swallowing the OFDI capsule OFDI, marking the region of interest, OFDI imaging, and removal of the OFDI capsule will take approximately 20 minutes
  The images obtained by the OFDI capsule will be compared to the images obtained by the clinical endoscopy and histology.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No